CLINICAL TRIAL: NCT04760925
Title: Single Arm, Open Label, Retrospective and Prospective Clinical Data Collection to Assess CascadeTM, Non-Occlusive Remodeling Net, in Providing Temporary Assistance for Coil Embolization of Intracranial Aneurysms
Brief Title: Cascade Clinical Data Collection Protocol
Status: Completed | Type: Observational
Sponsor: Perflow Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: CD0231
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CascadeTM, Non-Occlusive Remodeling Net — Temporary assistance device for coil embolization of intracranial aneurysms

SUMMARY:
This study is a multi-center, single arm, open label, retrospective and prospective clinical data collection of CascadeTM, Non-Occlusive Remodeling Net, in adults with intracranial aneurysms, demonstrating the effectiveness and safety of the CascadeTM in providing temporary assistance for coil embolization of intracranial aneurysms.

All consecutive eligible patients from all participating sites will be included in this clinical data collection. The relevant data of the coil embolization procedure will be collected via an eCRF system.

Peri procedural data on the coil embolization procedure as well as discharge, 30 days and at 3-6 months status will be collected.

ELIGIBILITY:
Patients must fulfill the following eligibility criteria to be included in the study:

1. Patient has been treated or planned to be treated with Cascade (Cascade device was opened).
2. Patient or patient's legally authorized representative or patient's family member (if approved by IEC) has signed and dated an Informed Consent Form (ICF), unless ICF is waived by local IEC.
3. Coil embolization procedure of intracranial aneurysm using temporary assisting device is initiated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were planned to undergo, or underwent coil embolization procedure of intracranial aneurysms assisted by the Cascade device
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2022-04-24 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint - Successful coil embolization of the target intracranial aneurysm assisted by Cascade device | During procedure
  Successful coil embolization of the target intracranial aneurysm assisted by Cascade device, without coil entanglement, protrusion or prolapse into the parent vessel at the end of the procedure, as evaluated angiographically by a central core-lab
Main Safety Endpoint - Incidence of Serious Adverse Device Effects (SADE) | within 30 days post procedure
  Serious adverse device effects (SADE) occurring within 30 days post procedure, including the following safety events:
  * Vessel damage related to the use of the study device that leads to dissection, perforation, hemorrhage or vasospasm.
  * Thromboembolic event related to the use of the study device.
  * Coil entanglement

SECONDARY OUTCOMES:
Secondary Efficacy Endpoint - Maintenance or improvement of aneurysm occlusion | 3-6 months post procedure
  Maintenance or improvement of aneurysm occlusion (evaluated angiographically by a central core-lab) using modified Raymond-Roy Classification (MRRC) at 3-6 months compared to the end of the procedure

OTHER OUTCOMES:
Other Safety Endpoint - Incidence of all Adverse Events | 30 days post procedure
  All adverse events experienced by enrolled patients within 30 days post coil embolization procedure, regardless of relatedness to the Cascade device or the coil embolization procedure

CONTACTS AND LOCATIONS:
Locations (7):
- UH St. Ivan Rilski, Sofia, Bulgaria
- Germany (2):
  - Medical Faculty of the Otto von Guericke University Magdeburg, Magdeburg
  - radprax MVZ GmbH, Solingen
- Sheba Medical Center, Tel Litwinsky, Israel
- Central Clinical Hospital of the MSWiA, Warsaw, Poland
- Spain (2):
  - Hospital Universitari De Bellvitge, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona